CLINICAL TRIAL: NCT00840294
Title: Randomized, Multi-Institution Trial of Ciprofloxacin Versus Observation for Men With an Elevated Prostate Specific Antigen (PSA)
Brief Title: Randomized Trial of Ciprofloxacin Versus Observation for Men With Elevated Prostate Specific Antigen (PSA)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Combination of futility analysis and poor accrual
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16368B
Record Dates: First submitted 2009-02-09; First posted 2009-02-10 (Estimated); Results first posted 2014-08-01 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Elevated Prostate Specific Antigen
Keywords: Men with Elevated PSA
MeSH Terms: interventions — Ciprofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Observation (No Intervention): Observation only for 2 weeks
- Antibiotic (Active Comparator): Ciprofloxacin 500 mg twice daily for 2 weeks
  Interventions: Drug: Ciprofloxacin

INTERVENTIONS:
Drug: Ciprofloxacin
  Other Names: Cipro
  Arms: Antibiotic

SUMMARY:
The purpose of this study is to assess the impact of an empiric course of antibiotics for men with an elevated prostate-specific antigen (PSA) level.

DETAILED DESCRIPTION:
Study Objectives:

Primary Objective: To assess the impact of ciprofloxacin on the change in PSA from baseline/randomization to prostate biopsy

Secondary Objective: To assess the impact of ciprofloxacin on the overall infectious complications following prostate biopsy

The impact of observation versus ciprofloxacin on PSA levels will be assessed by PSA change from baseline. The first PSA measurement will be at the study entry and randomization. The second PSA measurement will be immediately prior to prostate biopsy, which will occur 21-45 days following randomization.

ELIGIBILITY:
Inclusion Criteria:

* Men 18 yrs. or older
* An elevated PSA (>2.5 ng/ml) and normal digital rectal exam
* Have elected to proceed with a diagnostic 12-core prostate biopsy

Exclusion Criteria:

* Previous prostate biopsy
* History of prostate cancer
* Urinary tract infections or prostatitis within one year of study entry
* antibiotic use within one month prior to PSA level
* pyuria or bacteruria on urinalysis
* allergy to fluoroquinolones

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2009-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Eggener, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Observation | Antibiotic
Started | 42 | 43
Completed | 39 (These are the subjects included in the baseline, outcomes, and adverse events tables) | 38 (These are the subjects included in the baseline, outcomes, and adverse events tables)
Not Completed | 3 | 5
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Protocol Violation | 1 | 3
Not completed — Illness | 0 | 1

BASELINE CHARACTERISTICS:
Population: Subjects with complete data are included
Groups:
- Total: Total of all reporting groups
Arm/Group | Observation | Antibiotic | Total
Number analyzed (Participants) | 39 | 38 | 77
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 61.7 [55.5 to 66.7] | 60.4 [53.1 to 66.6] | 60.6 [53.1 to 66.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 39 | 38 | 77
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 23 | 26 | 49
  African-American | 12 | 10 | 22
  Other | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 39 | 38 | 77
PSA level [Mean (Full Range); unit: ng/mL] | 6.5 [2.4 to 17.4] | 7.6 [3.1 to 45.7] | 7.0 [2.4 to 45.7]

OUTCOME MEASURES:

1. Primary Outcome: Change in PSA Level From Baseline
Description: To assess the impact of ciprofloxacin on the change in PSA from baseline/randomization to prostate biopsy which occurs 21-45 days after randomization.
  Due to the skewness of the data, the log transformation was used and the outcome used was the log(PSA level post-treatment, at time of biopsy) - log(PSA level baseline).
Time Frame: At baseline and 21-45 days after randomization
Population: Subjects with complete data are included
Measure: Mean (Standard Deviation); unit: log ng/mL
Arm/Group | Observation | Antibiotic
Number analyzed (Participants) | 39 | 38
log ng/mL | -0.08 (0.39) | 0.005 (0.42)
Statistical Analysis 1: Comparison: Observation vs Antibiotic; Test type: Superiority or Other; p = 0.33, t-test, 2 sided

2. Secondary Outcome: Overall Infectious Complication Rate Following Prostate Biopsy
Description: To assess the impact of ciprofloxacin on the overall infectious complication rate following prostate biopsy
Time Frame: Within 24 hours of biopsy
Population: Subjects with complete data are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Observation | Antibiotic
Number analyzed (Participants) | 39 | 38
percentage of participants | 0 [0 to 9.0] | 2.6 [0.07 to 13.8]

ADVERSE EVENTS:
Time Frame: during the 2 weeks of study treatment
Description: Subjects with complete data are included.
Arm/Group | Observation | Antibiotic
Serious Adverse Events (participants affected / at risk) | 0/39 | 1/38
Other Adverse Events (participants affected / at risk) | 0/39 | 0/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Observation (N=39) | Antibiotic (N=38)
Sepsis (Infections and infestations) | 0 | 1

LIMITATIONS AND CAVEATS:
Early termination due to poor accrual and interim futility analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes